CLINICAL TRIAL: NCT01010360
Title: Identification of Celiac Ganglia for Endoscopic Ultrasound
Brief Title: Identification of Celiac Ganglia
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 0906-71
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Celiac Ganglia
Keywords: celiac ganglia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Computer-aided image recognition will improve the technique of endoscopic ultrasound-celiac plexus block/celiac plexus neurolysis (EUS-CPB/CPN) and improved pain relief.

DETAILED DESCRIPTION:
All subjects who are undergoing EUS will be eligible. Consecutive patients undergoing EUS will be invited to participate in this study. Subjects must be 18 years old or above at the time of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* all EUS patients

Exclusion Criteria:

* under 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: EUS patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia LeBlanc, MD, MPH, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States